CLINICAL TRIAL: NCT04479007
Title: Confocal Laser Endomicroscopy and Optical Coherence Tomography in Acute Respiratory Insufficiency
Brief Title: CLE and OCT in Acute Respiratory Insufficiency
Acronym: CLEOPATRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, Head of department of pulmonal endoscopy, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL61112.018.17
Record Dates: First submitted 2017-10-25; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Acute Respiratory Failure (Non Resolving)
Keywords: Confocal Laser Endomicroscopy; Optical coherence Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated patients: Critically ill patients of 18 years or older who receive invasive mechanical ventilation for acute respiratory failure and have an indication for an intervention in the airways.
  Interventions: Device: Probe based optical techniques

INTERVENTIONS:
Device: Probe based optical techniques — During the intervention of inspecting the airways, different segments of the alveolar compartment will be imaged by two different probe based (CLE and OCT).

SUMMARY:
Acute respiratory distress syndrome is a severe complication of critical illness. The diagnosis of ARDS is difficult, and it could be important to differentiate ARDS from other causes of acute respiratory failure. Innovative probe-based imaging techniques such as 'Confocal Laser Endomicroscopy' (CLE) and Optical Coherence Tomography (OCT) are high resolution optical techniques that, combined with conventional bronchoscopy, have been found to provide non-invasive, real-time near-histology information about the alveolar compartment in non ventilated non-critically ill patients.

DETAILED DESCRIPTION:
It is important to identify the underlying cause of respiratory failure, in order to determine the appropriate treatment. Histopathology would help treatment decisions, however is in the fast majority of this critically ill patient-group not available. CLE is enables near histology/microscopic analysis during bronchoscopy, by tissue illumination with a low-power laser. Optical Coherence Tomography is the optical equivalent of B-mode ultrasonography, that consists of a small rotating optical fibre. Both the CLE and OCT techniques are minimally invasive and little time consuming. Therefore different areas of the lung can be sequentially imaged. With this pilot study the investigators aim to describe normal alveolar areas and areas with abnormalities in critically ill patients with non resolving acute respiratory failure mandating a standard bronchoscopy or laryngoscopy with or without bronchoalveolar lavage.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care unit of academic medical center in Amsterdam
* Indication for a procedure to investigate the airways that can be combined with pCLE/OCT

Exclusion Criteria:

* Inability and willingness to provide informed consent by family-members
* Inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients mandating a procedure that includes inspection of the airways and can be combined with pCLE/OCT. Patients can only be included when the research physician decides they are eligible. (based on the heterogeneity of the disease and the suspected etiology).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-08-11 (Estimated); Study Completion 2020-08-11 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of various (diseased/non-diseased on HRCT-scan) alveolar compartments in mechanically ventilated patients | coss sectional (1 day)
  Percentage of successful imaging

SECONDARY OUTCOMES:
Comparison of pCLE/OCT to radiological patterns | cross sectional (1 day)
  Degree of similarity pCLE/OCT-imaging compared to HRCT
Comparison of pCLE/OCT with pathology | cross sectional (1 day)
  Degree of similarity between pCLE/OCT characteristics with pathology (in case available)

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Marcus J Schultz, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the data.